CLINICAL TRIAL: NCT05103969
Title: Multicenter Prospective Cohort of Tumors With Pole/D1 Mutation
Brief Title: Cohort of Tumors With POLE/D1 Mutation
Status: Recruiting | Type: Observational
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Other Study IDs: POLE COHORT
Record Dates: First submitted 2021-10-06; First posted 2021-11-02 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Tumors; POLE Exonuclease Domain Mutation; POLD1 Gene Mutation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blocks of tumor removed in the course of care fixed tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objective of this study is to identify and describe the clinico-biological and molecular characteristics of tumors with somatic POLE (Polymerase ɛ)/POLD1 mutation identified by molecular biology platforms for all stages and primary sites combined

DETAILED DESCRIPTION:
The identification of patients to be included will be done directly from the tumor genotyping platforms.

Indeed, they will be the direct source of the identification of all POLE (Polymerase ɛ) mutations.

The platforms will inform the project coordination unit of new cases of mutated cancers as well as the referent investigator, jointly they will be in charge of data entry.

The diagnostic and follow-up data of each patient will be collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Any tumor presenting a variant of the exonuclease domain of POLE (exons 9 to 14) classified as pathogenic by the project working group, including: the 4 hotspots of mutations described (codons 286 (P286R/H/L), 411 (V411L), 459 (S459F), 424 (L424/V/I), (2).
* Any tumor presenting a variant of the exonuclease domain of PolD1 (exons 8-12), classified as pathogenic by the project working group, including : C319Y(10).

Diagnosis made from the date of launch of the cohort and in the previous year

-Age ≥ 18 years

Exclusion Criteria:

* Tumor without POLE or POLD1 mutation
* Tumor with POLE mutation identified in research studies retrospective research
* Opposition of the patient to the registration of his data in the cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patient with a histologically proven tumor with a POLE or POLD1 mutation identified by molecular biology analysis, carried out within the framework of clinical practice in the platforms that have set up this research.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-10-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
To identify and describe the clinico-biological and molecular characteristics of tumors with somatic POLE/POLD1 mutation identified by molecular biology platforms for all stages and primary sites | October 2027
  Collection and description of clinical and histo-pathological data of tumors with POLE/POLD1 mutation
Molecular characterization of the identified POLE/POLD1 mutations | October 2027
  Molecular characterization of the identified POLE/POLD1 mutations and of the mutational profile associated with these mutations
Overall survival and response to treatments | October 2027
  Analysis of overall survival and response to treatments (chemotherapies, immunotherapies...)

SECONDARY OUTCOMES:
database and block librabry | October 2027
  Establishment of a database of somatic POLE variants Establishment of a block library of POLE mutated tumors

CONTACTS AND LOCATIONS:
Overall Officials: Rosine GUIMBAUD, PhD.MD, Principal Investigator — Fédération francophone de Cancérologie digestive
Locations (1):
- CHU -hopital Rangeuil, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided